CLINICAL TRIAL: NCT07194642
Title: Feasibility and Performance of Continuous Glucose Monitoring to Guide Computerized Insulin Infusion Therapy in Non-ICU Patients Receiving Corticosteroid Therapy and Specialized Nutrition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Principal Investigator, Andjela Drincic, Professor, University of Nebraska
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0144-25-FB
Record Dates: First submitted 2025-09-16; First posted 2025-09-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Inpatient patients meeting inclusion criteria and not exclusion criteria will be approached and consented by personnel listed in section I. Enrolled participants will be randomized to one of two arms:
  1. hybrid protocol originally developed by Faulds et al. integrating CGM with periodic POC-BG tests to monitor and ensure the ongoing accuracy of CGM measurements (available at http://www.covidindiabetes.org).
  2. standard care with hourly POC testing with blinded professional CGM for data analysis
Who Masked: Participant, Care Provider
Masking Description: he blinded CGM data will not be visible to the participant, nursing staff, or other care providers. The blinded CGM data will be used for data analysis following the completion of the participant's participation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Unblinded CGM (Other): Nursing staff will compare CGM and POC-BG readings every 1 to 2 hours using institutional blood glucose meters. Validated CII calculator will be utilized. Validation will be considered successful when two consecutive CGM readings were within 20% of the POC-BG when BG exceeded 100 mg/dL, or within 20 mg/dL if the POC-BG was below 100 mg/dL. The electronic health records (EHR) will utilize the CGM glucose value entered in the patient flowsheet row for comparison with POC-BG results using the published algorithm above to calculate, confirm, and record the success of the validation.
  - Ongoing validation phase for the sustained use of CGM. After the initial CGM validation, POC-BG checks and the CGM validation will be reduced to every 6 hours, and CII titration in the interim was guided by CGM values until the next POC-BG assessment.
  Interventions: Other: Dexcom G7 CGM
- Blinded CGM (Other): After CGMs are placed (on the abdomen in all participants) and have completed their warm-up period, the nursing staff will proceed with standard of care POC finger sticks. The blinded CGM data will not be visible to the participant, nursing staff, or other care providers. The blinded CGM data will be used for data analysis following the completion of the participant's participation.
  Interventions: Other: Dexcom G7 CGM

INTERVENTIONS:
Other: Dexcom G7 CGM — The Dexcom G7 is a continuous glucose monitor, FDA 510K cleared (K213919) for people with diabetes. Worn for 10 days at a time, the device monitors the glucose levels of interstitial fluid and, via bluetooth, transmits data every 5 minutes to a receiver.

SUMMARY:
The objective of this pilot study is to assess the feasibility and performance of real-time CGM for titrating CII via: (1) evaluation of CGM glucose accuracy in oncology and post-transplant population receiving IV insulin therapy, and (2) assessing both nursing acceptance/convenience and patient satisfaction with CGM use. A randomized prospective trial model will be used comparing glucose control (glucometrics hypoglycemia), patient experience and nursing satisfaction in cancer patients receiving IV insulin therapy where monitoring is done via: a) hybrid protocol originally developed by Faulds et al. integrating CGM with periodic POC-BG tests to monitor and ensure the ongoing accuracy of CGM measurements (available at http://www.covidindiabetes.org). b) standard care with hourly POC testing and blinded professional CGM.Inclusion criteria: Eligible patients include oncology and post-transplant patients receiving IV insulin therapy while on corticosteroid treatment and receiving specialized nutrition. Exclusion criteria: medically instable patients receiving pressor therapy and ICU level of care. Outcome evaluation; Patients' characteristics were collected through the EHR. Glucometrics will be collected throughout the study to include mean BS, % in range ( 80-180) , patient day hypoglycemia , patient stay hypoglycemia . Nursing surveys: Survey will be provided for nurses to assess nursing burden, acceptability. Nurses will complete a survey before starting the project and again after being involved in the initial and ongoing validation phases of CGM at the end of the project. The purpose is to report their convenience with using CGM and their preferred glucose monitoring method, which included POC arterial blood, POC finger sticks, and CGM. Nursing surveys will be administrated electronically to nursing staff and the results will be uploaded automatically. Patient survey: Patients will be approached by the team members to inquire about the willingness to provide feedback. The questionnaire will assess their experiences of care with CGM (options: very good, good, fair, poor), glucose check without pain and disruptions of sleep (yes/no), and overall confidence of care with CGM process (very confident, quite confident, somewhat confident, little confident). Patient surveys will handed out by the team members, and the results were subsequently entered into database (See both nursing and patient surveys in Supplementary Material.)

DETAILED DESCRIPTION:
The objective of this pilot study is to assess the feasibility and performance of real-time CGM for titrating Continuous Insulin Infusion Therapy (CII) via: (1) evaluation of CGM glucose accuracy in oncology and post-transplant population receiving IV insulin therapy, and (2) assessing both nursing acceptance/convenience and patient satisfaction with CGM use. (3) Background and Rationale

Managing blood glucose in the hospital is challenging but important. Hypoglycemia and hyperglycemia have been associated with increased length of stay, decreased wound healing, and mortality. For patients experiencing severe hyperglycemia and for those with rapidly changing insulin requirement, insulin infusion therapy is considered a mainstay of hospital management. The short half-life of intravenous insulin allows for precise titration of insulin drip that is facilitated by frequent glucose monitoring. However CII therapy also poses unique challenges. Safe administration of insulin by this route is very labor intensive for the nursing staff. This is particularly true for patients receiving insulin drips on the general floor and step down unit where nursing/patient ratios are typically 1-4 to 1-6 .

Placing a CGM sensor on these patients would provide nursing staff with the ability to monitor blood glucose levels with minimal patient disruption for finger stick glucose checks. The use of CGM is endorsed by Endocrine Society's 2022 Guidelines to effectively achieve glycemic targets and reduce hypoglycemia in hospitalized patients. Adjunctive use of CGM in addition to POC testing has been described as safe and effective for patients receiving insulin drips.

In addition, utilizing insulin drips for days on, is burdensome for the patient due to hourly finger sticks and disruption of sleep and impaired wellbeing associated with the process. Evidence demonstrates decreasing sleep disruptions may reduce delirium, hypertension, and mortality and improve the overall patient experience. Current standard of care requires that patients receiving insulin infusions receives POC monitoring every 1-2 hours, day or night, resulting in significant pain associated with PPC testing and the need to wake patients up during their sleep. With the adjunctive use of CGM monitoring POC testing would be reduced to every 6 hours.

Lastly, safety is an important consideration. Hypoglycemia is a common complication of insulin therapy even with close monitoring. In our institution, last year there were 210 hypoglycemic events were recorded for patients receiving insulin infusions (~ 8.6% of patients on insulin drips). The causes are multifactorial, with significant contribution of those related to algorithm adjustment, however failure to keep with hourly POC due to time constraints and logistical barriers in workflow contributed.

A 2018 study found the average marginal cost for an inpatient stay with a hypoglycemic adverse event was $4,312 per event. This increase in cost is related to an increase in average length of stay, an increase of 38.9% in total charges, increase in likelihood of requiring skilled nursing care post discharge, and a 7% increase of in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age >19 years old
* Patients with diabetes or stress induced hyperglycemia requiring continuous insulin infusion therapy, with anticipated duration of this therapy being > 24 hours. Specifically, we will include
* Patients with Type 2 diabetes; or if not previously diagnosed as having diabetes, HbA1c >7.0% (laboratory-measured at or since hospital admission or within prior 3-months).
* Type 1 diabetes, as well as atypical forms of diabetes (including pancreatectomy and pancreatitis) and
* Stress hyperglycemia defined as at least 1 blood glucose measurement >180 mg/dL since admission in a patient without history of diabetes, if CII is indicated per treating physician
* Insulin drip (CII) already initiated since admission or planned to be initiated
* Non-critical hospitalization with expected duration of CII > 24 hours at time of randomization
* Oncology and post-transplant population receiving IV insulin therapy

Exclusion Criteria:

* Inability to provide written consent
* Medically unstable patients receiving pressor therapy and ICU level of care.
* Patients transferred from ICU with an expected requirement for CII > 24 hours on a non-ICU floor are eligible)
* For women of childbearing potential: currently pregnant or breastfeeding
* Hypoxia (O2 saturation < 90 %) present at time of potential enrollment
* Hemoglobin < 7 mg/dL;
* Anasarca present at time of potential enrollment
* Use of hydroxyurea or high dose acetaminophen use of >4g daily as those are substances known to interfere with CGM system.
* eGFR < 20 mL/min or dialysis being received or planned
* Known allergy to medical grade adhesives or a skin condition that may impact CGM performance per investigator discretion
* Admission for Diabetic ketoacidosis or hyperosmolar hyperglycemic state

Nurse Participants:

* Adults aged 19 and older involved in the routine care of the patient participants
* Adequate proficiency to understand and provide informed consent in English

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority for TIR (Time in Range) | 12 Months
  Participant characteristics will be collected through the EHR. Descriptive analyses will be conducted to summarize patient characteristics, POC-BG, CGM data and survey data.

REFERENCES:
- [Background] Tian T, Aaron RE, Yeung AM, Huang J, Drincic A, Seley JJ, Wallia A, Gilbert G, Spanakis EK, Masharani U, Faulds E, Hirsch IB, Dawood GE, Espinoza JC, Mendez CE, Kerr D, Klonoff DC. Use of Continuous Glucose Monitors in the Hospital: The Diabetes Technology Society Hospital Meeting Report 2023. J Diabetes Sci Technol. 2023 Sep;17(5):1392-1418. doi: 10.1177/19322968231186575. Epub 2023 Aug 9. PMID 37559371
- [Background] Nair BG, Dellinger EP, Flum DR, Rooke GA, Hirsch IB. A Pilot Study of the Feasibility and Accuracy of Inpatient Continuous Glucose Monitoring. Diabetes Care. 2020 Nov;43(11):e168-e169. doi: 10.2337/dc20-0670. Epub 2020 May 11. No abstract available. PMID 32393587
- [Background] Dillmann C, Amoura L, Fall Mostaine F, Coste A, Bounyar L, Kessler L. Feasibility of Real-Time Continuous Glucose Monitoring Telemetry System in an Inpatient Diabetes Unit: A Pilot Study. J Diabetes Sci Technol. 2022 Jul;16(4):955-961. doi: 10.1177/1932296821994586. Epub 2021 Mar 4. PMID 33660531
- [Background] Curkendall SM, Natoli JL, Alexander CM, Nathanson BH, Haidar T, Dubois RW. Economic and clinical impact of inpatient diabetic hypoglycemia. Endocr Pract. 2009 May-Jun;15(4):302-12. doi: 10.4158/EP08343.OR. PMID 19502209
- [Background] Stewart NH, Arora VM. Sleep in Hospitalized Older Adults. Sleep Med Clin. 2018 Mar;13(1):127-135. doi: 10.1016/j.jsmc.2017.09.012. Epub 2017 Nov 10. PMID 29412979
- [Background] Clarke WL, Cox D, Gonder-Frederick LA, Carter W, Pohl SL. Evaluating clinical accuracy of systems for self-monitoring of blood glucose. Diabetes Care. 1987 Sep-Oct;10(5):622-8. doi: 10.2337/diacare.10.5.622. PMID 3677983
- [Background] Faulds ER, Jones L, McNett M, Smetana KS, May CC, Sumner L, Buschur E, Exline M, Ringel MD, Dungan K. Facilitators and Barriers to Nursing Implementation of Continuous Glucose Monitoring (CGM) in Critically Ill Patients With COVID-19. Endocr Pract. 2021 Apr;27(4):354-361. doi: 10.1016/j.eprac.2021.01.011. Epub 2021 Jan 27. PMID 33515756
- [Background] Faulds ER, Boutsicaris A, Sumner L, Jones L, McNett M, Smetana KS, May CC, Buschur E, Exline MC, Ringel MD, Dungan K. Use of Continuous Glucose Monitor in Critically Ill COVID-19 Patients Requiring Insulin Infusion: An Observational Study. J Clin Endocrinol Metab. 2021 Sep 27;106(10):e4007-e4016. doi: 10.1210/clinem/dgab409. PMID 34100545
- [Background] Ang L, Lin YK, Schroeder LF, Huang Y, DeGeorge CA, Arnold P, Akanbi F, Knotts S, DuBois E, Desbrough N, Qu Y, Freeman R, Esfandiari NH, Pop-Busui R, Gianchandani R. Feasibility and Performance of Continuous Glucose Monitoring to Guide Computerized Insulin Infusion Therapy in Cardiovascular Intensive Care Unit. J Diabetes Sci Technol. 2024 May;18(3):562-569. doi: 10.1177/19322968241241005. Epub 2024 Apr 2. PMID 38563491